CLINICAL TRIAL: NCT05644431
Title: A Prospective Clinicobiological Cohort Study Aiming to Decipher Tumor Immune Microenvironment Evolution Under Standard Chemotherapy in Localized and Resectable Gastric and Gastroesophageal Junctional Adenocarcinomas
Brief Title: GastrOesophageal Tumor, Immune Microenvionnment (GOTIM)
Acronym: GOTIM
Status: Recruiting | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: ET22-201
Record Dates: First submitted 2022-11-21; First posted 2022-12-09 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: GastroEsophageal Cancer
Keywords: junctional adenocarcinomas; immune microenvironment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor samples to be collected include:
  1. Mandatory archival FFPE tumor block from initial diagnosis biopsy.
  2. Mandatory fresh tumor samples performed before neoadjuvant CT and collected during gastroscopy.
  3. Mandatory FFPE tumor samples from surgery specimen and lymph nodes collected during surgery.
  4. Optional FFPE tumor block from biopsy or surgery in case of relapse.
  Blood samples to be collected include:
  1. At D1 pre-dose of neoadjuvant CT treatment
  2. End of neoadjuvant treatment i.e. within at 1 month after the last neoadjuvant treatment
  3. At surgery (within 2 days before or after surgery)
  4. At M3, M6, M9, M12, M15, M19, M21, M24, M30, M36
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastric and gastroesophageal junctional adenocarcinomas: Patient under standard chemotherapy in localized and resectable gastric and gastroesophageal junctional adenocarcinomas

SUMMARY:
This trial is a prospective, monocentric, non-therapeutic, interventional cohort study aiming to decipher the immune TME through standard neoadjuvant CT in resectable G/GEJ adenocarcinomas. This study will also longitudinally monitor MRD during neoadjuvant and adjuvant therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient > 18 years of age on day of signing informed consent.
* Histologically proven non-metastatic resectable gastric and gastroesophageal junction adenocarcinoma, Stage IB to III to be treated with standard neoadjuvant treatment.
* Surgery of primary tumor to be done at Centre Léon Bérard.
* Availability of archival FFPE tumor block from initial diagnosis with at least 20% of tumor cells.
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0, 1 or 2.
* Patient should understand, sign, and date the written voluntary informed consent form at the screening visit prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedures as per protocol.
* Patients must be covered by a medical insurance.

Exclusion Criteria:

* Any condition contraindicated with blood sampling procedures required by the protocol.
* Known additional malignancy that is progressing or requires active treatment. Exceptions include adequately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer
* Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure.
* Pregnant or breast-feeding woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with localised non-metastatic operable gastric and oeasogatric junction adenocarcinoma, stage IB à III, treated with standard neoadjuvant therapy and by surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-07-19 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Describe Gastric and Gastroesophageal immunological tumor microenvironment | At least 36 months following inclusion
  Spatial, spectral cytometry, and transcriptomic analyses

SECONDARY OUTCOMES:
Understand the evolution of the immune tumor microenvironment and its spatial structuration through standard neoadjuvant chemotherapy. | At least 36 months following inclusion
Characterize the evolution of the immune tumor environment profiles and organization between responder and non-responder patients under standard neoadjuvant treatment. | At least 36 months following inclusion
Characterize the immune profile in lymph nodes after surgery (lymphadenectomy) between responder and non-responder patients to neoadjuvant under standard neoadjuvant treatment. | At least 36 months following inclusion
Assess the phenotype and functions of circulating immunes cells | At least 36 months following inclusion
Perform integrative analysis combining spatial, molecular, single cell RNAseq, and spectral flow cytometry analysis on the immunological tumor environment in matched tumor tissues longitudinally | At least 36 months following inclusion

OTHER OUTCOMES:
evaluate in patient-derived tumor fragment (ex vivo platform of Centre Léon Bérard), the impact of immune checkpoint inhibitors (ICI) selected from our previous data in order to develop and improve therapeutic strategy | At least 36 months following inclusion
assess MRD using liquid biopsies over standard neoadjuvant and adjuvant treatment. | At least 36 months following inclusion
assess the correlation between ctDNA analysis and i) patient clinical outcome and ii) current prognostic factors (for instance TNM stage with ypTN stage in gastric and oesogastric junction carcinomas). | At least 36 months following inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Clélia COUTZAC, MD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard, Lyon, France